CLINICAL TRIAL: NCT00003292
Title: S9624: Phase II Study of Ifosfamide in Patients With Aggressive Meningeal Tumors
Brief Title: S9624 Ifosfamide in Treating Patients With Meningeal Tumors
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: lack of accrual
Sponsor: SWOG Cancer Research Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH); Eastern Cooperative Oncology Group (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000066225; S9624 (Other: SWOG); U10CA032102 (NIH)
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Last update posted 2013-11-08 (Estimated); Status verified 2013-11

CONDITIONS: Chondrosarcoma; Adult Fibrosarcoma; Adult Leiomyosarcoma; Adult Rhabdomyosarcoma; Adult Malignant Meningioma; Adult Brain Malignant Hemangiopericytoma
MeSH Terms: conditions — Chondrosarcoma; Fibrosarcoma; Leiomyosarcoma; Rhabdomyosarcoma; Meningioma | interventions — Ifosfamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- ifosfamide (Experimental): ifosfamide
  Interventions: Drug: ifosfamide

INTERVENTIONS:
Drug: ifosfamide

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase II trial to study the effectiveness of ifosfamide in treating patients with meningeal tumors that have recurred or that cannot be removed surgically.

DETAILED DESCRIPTION:
OBJECTIVES:

* Estimate failure free survival, overall survival, and response in patients with residual or recurrent/progressive aggressive meningeal tumors (malignant meningioma, hemangiopericytoma, and primary nervous system sarcoma) treated with ifosfamide.
* Evaluate toxicities of ifosfamide in this patient population.

OUTLINE: All patients receive ifosfamide IV continuously over 72 hours on days 1-3 of each 21 day treatment course. Patients are evaluated for response/progression after every 2 courses. Patients with stable disease receive up to 8 courses of therapy. Treatment continues in the absence of disease progression or unacceptable toxicity.

Patients are followed every 3 months for 1 year, then every 6 months thereafter.

PROJECTED ACCRUAL: Approximately 35 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically proven recurrent or unresectable:
* Malignant meningioma
* Intracranial hemangiopericytoma
* Primary central nervous system sarcoma, including:
* Fibrosarcoma
* Rhabdomyosarcoma
* Chondrosarcoma
* Leiomyosarcoma
* Measurable or evaluable disease on CT or MRI scan
* Persistent disease following biopsy or incomplete resection OR
* Recurrent disease following complete resection
* No benign meningioma
* No prior or current systemic sarcoma

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* SWOG 0-2

Life expectancy:

* Not specified

Hematopoietic:

* WBC at least 3,000/mm^3
* Absolute granulocyte count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3

Hepatic:

* Not specified

Renal:

* Creatinine no greater than 2.0 mg/dL

Cardiovascular:

* No myocardial infarction within the past 3 months
* No active angina
* No unstable heart rhythms
* No congestive heart failure

Other:

* HIV negative
* No allergy to study drugs
* No serious concurrent medical or psychiatric illness
* No uncontrolled peptic ulcer disease
* No prior malignancy within past 5 years except adequately treated:
* Basal or squamous cell carcinoma of the skin
* Carcinoma in situ of the cervix
* Not pregnant or nursing
* Effective contraception required of fertile patients

PRIOR CONCURRENT THERAPY:

* Recovered from toxic effects of prior therapy and/or from postoperative complications

Biologic therapy:

* Not specified

Chemotherapy:

* No prior ifosfamide
* No other concurrent chemotherapy

Endocrine therapy:

* No concurrent hormonal therapy (except estrogen replacement therapy)
* Corticosteroids allowed if dose is stable or decreasing

Radiotherapy:

* At least 4 weeks since prior radiotherapy
* Progressive disease following radiation required
* No concurrent radiotherapy

Surgery:

* See Disease Characteristics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 1998-07; Primary Completion 2004-01 (Actual); Study Completion 2004-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Leslie McAllister, MD, Study Chair — Neurological Clinic; Lynn G. Feun, MD, Study Chair — University of Miami Sylvester Comprehensive Cancer Center
Locations (70):
- United States (65):
  - CCOP - Scottsdale Oncology Program, Scottsdale, Arizona
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Veterans Affairs Medical Center - Palo Alto, Palo Alto, California
  - Stanford University Medical Center, Stanford, California
  - CCOP - Colorado Cancer Research Program, Incorporated, Denver, Colorado
  - CCOP - Christiana Care Health Services, Newark, Delaware
  - Veterans Affairs Medical Center - Gainesville, Gainesville, Florida
  - H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - Veterans Affairs Medical Center - Tampa (Haley), Tampa, Florida
  - Emory University Hospital - Atlanta, Atlanta, Georgia
  - Veterans Affairs Medical Center - Atlanta (Decatur), Decatur, Georgia
  - CCOP - Central Illinois, Decatur, Illinois
  - CCOP - Evanston, Evanston, Illinois
  - CCOP - Illinois Oncology Research Association, Peoria, Illinois
  - CCOP - Carle Cancer Center, Urbana, Illinois
  - Indiana University Cancer Center, Indianapolis, Indiana
  - Veterans Affairs Medical Center - Indianapolis (Roudebush), Indianapolis, Indiana
  - CCOP - Cedar Rapids Oncology Project, Cedar Rapids, Iowa
  - CCOP - Iowa Oncology Research Association, Des Moines, Iowa
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - Mercy Medical Center, Des Moines, Iowa
  - Iowa Lutheran Hospital, Des Moines, Iowa
  - MBCCOP - LSU Health Sciences Center, New Orleans, Louisiana
  - CCOP - Ochsner, New Orleans, Louisiana
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - Tuft-New England Medical Center, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - CCOP - Michigan Cancer Research Consortium, Ann Arbor, Michigan
  - CCOP - Kalamazoo, Kalamazoo, Michigan
  - Veterans Affairs Medical Center - Minneapolis, Minneapolis, Minnesota
  - University of Minnesota Cancer Center, Minneapolis, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - CCOP - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - Alegent Health-Midlands Community Hospital, Papillion, Nebraska
  - CCOP - Southern Nevada Cancer Research Foundation, Las Vegas, Nevada
  - Veterans Affairs Medical Center - East Orange, East Orange, New Jersey
  - CCOP - Northern New Jersey, Hackensack, New Jersey
  - Cancer Institute of New Jersey, New Brunswick, New Jersey
  - MBCCOP - University of New Mexico HSC, Albuquerque, New Mexico
  - Veterans Affairs Medical Center - Brooklyn, Brooklyn, New York
  - Veterans Affairs Medical Center - New York, New York, New York
  - NYU School of Medicine's Kaplan Comprehensive Cancer Center, New York, New York
  - James P. Wilmot Cancer Center, Rochester, New York
  - Albert Einstein Clinical Cancer Center, The Bronx, New York
  - Veterans Affairs Medical Center - Fargo, Fargo, North Dakota
  - CCOP - Merit Care Hospital, Fargo, North Dakota
  - Ireland Cancer Center, Cleveland, Ohio
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - CCOP - Columbus, Columbus, Ohio
  - CCOP - Oklahoma, Tulsa, Oklahoma
  - CCOP - Geisinger Clinic and Medical Center, Danville, Pennsylvania
  - Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Drexel University Hospital, Philadelphia, Pennsylvania
  - Kimmel Cancer Center of Thomas Jefferson University - Philadelphia, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - University of Pittsburgh Cancer Institute, Pittsburgh, Pennsylvania
  - Veterans Affairs Medical Center - Pittsburgh, Pittsburgh, Pennsylvania
  - CCOP - MainLine Health, Wynnewood, Pennsylvania
  - CCOP - Sioux Community Cancer Consortium, Sioux Falls, South Dakota
  - CCOP - St. Vincent Hospital Cancer Center, Green Bay, Green Bay, Wisconsin
  - Veterans Affairs Medical Center - Madison, Madison, Wisconsin
  - University of Wisconsin Comprehensive Cancer Center, Madison, Wisconsin
  - CCOP - Marshfield Medical Research and Education Foundation, Marshfield, Wisconsin
  - Medical College of Wisconsin Cancer Center, Milwaukee, Wisconsin
  - Veterans Affairs Medical Center - Milwaukee (Zablocki), Milwaukee, Wisconsin
- Westmead Hospital, Westmead, New South Wales, Australia
- Instituto de Enfermedades Neoplasicas, Lima, Peru
- Puerto Rico (3):
  - MBCCOP - San Juan, San Juan
  - Veterans Affairs Medical Center - San Juan, San Juan
  - San Juan City Hospital, San Juan